CLINICAL TRIAL: NCT06528353
Title: SCREEN-HPV: Blood Biomarkers Based Screening for HPV-driven OPC
Brief Title: Blood Biomarkers Based Screening for HPV-driven OPC
Acronym: SCREEN-HPV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ORL 16
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Anal Cancer; Human Papilloma Virus
Keywords: HPV-induced cancer; Head and Neck Cancers; virology; serology; secondary cancer prevention
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): For the first 500 participants enrolled, one additional blood sample will be drawn in DNA-free tubes for HPV ctDNA analysis. As we expect to have around 1% seropositive cases, most of these 500 samples will be seronegative and will constitute our control group. These controls will be tested for HPV ctDNA to confirm that seronegative participants are also HPV ctDNA-negative
  Interventions: Diagnostic Test: HPV16-E6 serology and HPV ctDNA
- Experimental Group (Experimental): Individuals who are seropositive for HPV16-E6 will be contacted to propose the participation in the second part of the study and benefit from specific assessment and monitoring for 5 years (HPV ctDNA testing, regular clinical examinations of the head & neck and anal-genital regions, imaging if needed).
  Interventions: Diagnostic Test: HPV16-E6 serology and HPV ctDNA

INTERVENTIONS:
Diagnostic Test: HPV16-E6 serology and HPV ctDNA — In the event of a malignant lesion identified on clinical examination and/or imaging, treatment will be performed according to the standard of care. In the absence of any suspicious lesion, but in the event of HPV ctDNA positivity, prophylactic surgery of the tonsils and base of the tongue (the vast majority of HPV-related OPC develop in these regions) will be proposed to the patient, given the high risk of OPC. In case of refusal of this prophylactic surgery, close clinical and imaging monitoring will be performed.
  Surgical specimens will be analyzed to confirm or not the presence of HPV-driven OPC and HPV ctDNA will be measured post-operatively to ensure disease clearance.

SUMMARY:
The objective of our study is to demonstrate that it is possible to detect and treat human papilloma virus (HPV)-related oropharyngeal cancers (OPC) early using simple blood tests. The success of this strategy will be evaluated by the number of participants positive for both HPV16-E6 serology and HPV circulating tumor DNA (ctDNA) whose early management has allowed the detection of a cancerous lesion and/or whose HPV ctDNA results have normalized after surgical intervention. If this study is conclusive, it could pave the way for the implementation of a national screening strategy for HPV-related OPC.

DETAILED DESCRIPTION:
OPC caused by HPV are the most common head and neck cancers and are expected to increase in the future, especially since HPV vaccines are not widely used. Currently, there are no screening strategy available for these cancers, but developing such approaches could enable the earlier management of patients and thus improve prognosis while reducing treatment related toxicities.

Traditional screening methods like imaging or examination are not effective for OPC because early lesions are undetectable. However, studies suggest that using certain blood tests to detect HPV-related OPC early might be efficient:

* Antibodies directed against a specific protein of HPV called HPV16-E6 are present in most cases of HPV-related OPC and it has been shown that they can, be detected several years before the cancer diagnosis.
* HPV ctDNA can be found in the blood of almost all patients with HPV-related cancers. After treatment, HPV ctDNA can detect relapses before they are visible on imaging tests (microscopic disease) We propose to test the use of these two blood tests to identify individuals at high risk of developing OPC and offer them appropriate medical follow-up. HPV16-E6 serology will be conducted on 10,000 men over 50 years of age without symptoms who have consented to participate in the project. These participants will be included during routine visits to the biomedical analysis laboratory.

Individuals positive for HPV16-E6 test will be contacted (approximately 100 participants). They will be offered to continue the study to receive an initial assessment and regular monitoring for 5 years (HPV ctDNA test, regular clinical examinations, imaging examinations if needed). In case of identification of suspicious lesions, appropriate management will be proposed according to the standard recommendations. If no lesion is detected but HPV ctDNA remains positive, preventive surgery may be considered.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥50 years from the general population
* Man
* No previous history of HPV-driven cancer or head neck cancer
* Willingness to complete follow up visits

Exclusion Criteria:

* Aged < 50 years
* Woman
* History of HPV-driven cancer or head and neck cancer
* Psychiatric conditions
* Inability to complete follow up visits
* Severe medical condition (life expectancy <5 years)
* Previous prophylactic HPV vaccination

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2032-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Early identification of HPV-driven OPC lesions | 3 months following last prophylactic surgery
  The efficacy of this stepwise, biomarker-based screening approach to identify and treat early HPV-driven OPC lesions in asymptomatic individuals at high risk is determined by the number (and percentage) of participants who are positive for both HPV EA serology and HPV ctDNA, AND who have a successful identification of a tumor lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Haïtham Mirghani, Principal Investigator — APHP

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.